CLINICAL TRIAL: NCT06523868
Title: Evaluation of Multi-Cancer Early Detection Testing in a High-Risk Military Population: The Sentinel Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Principal Investigator, Elizabeth ODonnell, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 24-277
Record Dates: First submitted 2024-07-23; First posted 2024-07-26 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-03

CONDITIONS: Cancer Diagnosis
Keywords: Cancer Diagnosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Galleri MCED Test (Experimental): Enrolled participants will complete:
  * Baseline visit with blood draw and questionnaires
  * Return of study test result
  * Online post-test questionnaire
  * For a positive result, diagnostic work-up could include clinic visits, biopsy, surgery, imaging assessments such as ultrasound, Computed Tomography (CT) scans, or Magnetic Resonance Imaging (MRI) scans. If no cancer is found upon work up, a repeat MCED test may be ordered at the discretion of the principle investigator for up to 1 year from the initial MCED blood test.
  * Follow-up for a negative MCED blood test could include a repeat test ordered by the principle investigator for up to 1 year from the initial MCED test or a survey or phone call by study staff approximately 1 year after the initial MCED blood test.
  * Online post-diagnostic questionnaire.
  Interventions: Other: GRAIL Galleri

INTERVENTIONS:
Other: GRAIL Galleri — A multi-cancer early detection (MCED) blood test.

SUMMARY:
The purpose of this research study is to evaluate the possible benefits of an investigational, but commercially available Galleri multi-cancer early detection (MCED) blood test which is designed to detect many types of cancer early in veterans who have served in the military in active duty.

The name of the screening blood test being studied is:

-GRAIL Galleri MCED test

DETAILED DESCRIPTION:
This research study aims to assess the performance of the Galleri multi-cancer early detection (MCED) screening test in a military population and to compare the number and types of cancers diagnosed using MCED testing versus standard of care. This research study will give doctors and participants results of Galleri® blood tests which is designed to detect many types of cancer.

The research study procedures including screening for eligibility, blood draws, questionnaires, and clinic visits.

Participation in this research study is expected to last for up to 1 year.

It is expected that about 1,500 people will take part in this research study.

The Department of Defense (DoD) is funding this study.

ELIGIBILITY:
Inclusion Criteria:

* Active-duty or National Guard/Reserves military service for eight or more years
* Age ≥ 45
* Received care at a VA facility within past 5 years
* Able to sign informed consent
* Willingness to travel to Dana-Farber Cancer Institute in Boston, MA, for diagnostic testing if screening test indicates possible malignancy

Exclusion Criteria:

* Individuals diagnosed with invasive malignancy within 3 years of enrollment (non- melanoma skin cancer is acceptable)
* Individuals with evidence of symptomatic or active cancer requiring therapeutic intervention at the time of participation (hormone therapy for breast/prostate cancer is acceptable)
* Individuals in the process of being evaluated for a clinical suspicion of cancer

Min Age: 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1500 (Estimated)
Dates: Start 2025-03-31 (Actual); Primary Completion 2027-09-30 (Estimated); Study Completion 2028-09-30 (Estimated)

PRIMARY OUTCOMES:
Positive predictive value at 12 Months | At 12 months
  Positive predictive value is defined as the proportion of participants with cancer diagnosis out of all participants with "signal detected" on GRAIL Galleri MCED test results.
Negative predictive value at 12 Months | At 12 months
  Negative predictive value is defined as the proportion of participants with no cancer diagnosis out of all participants with "signal not detected" on GRAIL Galleri MCED test results.
Specificity Rate at 12 Months | At 12 months
  Specificity is defined as the proportion of participants with "signal not detected" results out of all participants with no cancer diagnosis on GRAIL Galleri MCED test results.
Yield Rate at 12 Months | At 12 months
  Yield rate is defined as the proportion of participants with "signal detected" out of all participants tested on GRAIL Galleri MCED test.
Number of Participants Needed to Screen at 12 months | At 12 months
  Number Needed to Screen (NNS) is defined as the number of participants screened to detect a diagnosis of invasive cancer on the GRAIL Galleri MCED test.

SECONDARY OUTCOMES:
Cancer Detection Rate Comparison | Up to 12 months
  Descriptive statistics will be used to summarize the number and types of cancers diagnosed by GRAIL Galleri MCED testing compared to Standard of Care (SOC) in matched population from the VA (separate IRB protocol).
Stage of Invasive Cancer Diagnosis Comparison | Up to 12 months
  Descriptive statistics will be used to summarize the stages of invasive cancer that are diagnosed by GRAIL Galleri MCED testing assessed by medical record review compared to Standard of Care (SOC) in matched population from the VA (separate IRB protocol).
Change in PROMIS Anxiety Short Form Score | Baseline to 12 months
  Changes in anxiety following the GRAIL Galleri MCED test result and assessed by the Patient-Reported Outcome Measurement Information System (PROMIS) Emotional Distress Anxiety - Short Form 6a, which is a 6 item survey that is rated on a 5-point Likert scale with answers ranging from "Never" to "Always". The range of scoring is from 6 to 30 with higher scores indicating greater severity of anxiety.
Change in PROMIS Global Health Score | Baseline to 12 months
  Changes in health-related quality of life following the GRAIL Galleri MCED test result and assessed by PROMIS Scale v1.2 - Global Health, a 10 item survey that is rated on a 5-point Likert scale with answers ranging from "Excellent/Completely/Never/None" to "Poor/Not at all/Always/Very Severe" and includes a pain average question rated on a scale of 0 "No Pain" to 10 "Worst Pain Imaginable." The range of scoring is from 9 to 45 with higher scores indicating higher quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth ODonnell, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (1):
- Dana-Farber Cancer Institute, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Belfer Office for Dana-Farber Innovations (BODFI) at innovation@dfci.harvard.edu